CLINICAL TRIAL: NCT05742971
Title: Virtual Reality; the Effect on Pain Reduction During an External Version, a Randomised Controlled Trial
Brief Title: Virtual Reality; the Effect on Pain Reduction During an External Version.
Acronym: VIREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NL-71484.096.19
Record Dates: First submitted 2023-02-09; First posted 2023-02-24 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2023-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study population will be randomly divided into the intervention group (VR-group) or the standard care group. The intervention group can choose for an immersive guided relaxation VR experience or an interactive VR experience during the external version additional to the usual standard care. The participants randomised to the standard care group receive the usual standard care given during external version.
Who Masked: Investigator
Masking Description: The study population will be randomly divided into the intervention group (VR-group) or the standard care group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): The intervention group can choose for an immersive guided relaxation VR experience or an interactive VR experience during the external version Immediately after the external version, a pain measurement is taken with regard to the pain during the ECV by means of the NRS score. After the ECV procedure, participants of the VR-group receive a structured questionnaire in which tolerability, feasibility and satisfaction of VR use is evaluated.
  Interventions: Device: Virtual reality intervention performed through the Oculuc Go VR glasses
- Standard care group (No Intervention): The participants randomised to the standard care group receive the usual standard care given during external version.Immediately after the external version, a pain measurement is taken with regard to the pain during the ECV by means of the NRS score.

INTERVENTIONS:
Device: Virtual reality intervention performed through the Oculuc Go VR glasses — The participants randomised into this group are offered a VR intervention during the external version for 5-10 minutes in addition to the standard care of an ECV. The VR is performed through the Oculus Go VR glasses. These women can choose for an immersive guided relaxation VR experience or an interactive VR experience (see descriptions below). The ECV expert executing the ECV will register immediately after the ECV which option the patients has chosen. Immediately after the external version, a pain measurement is taken with regard to the pain during the ECV by means of the NRS score. After the ECV procedure, participants of the VR-group receive a structured questionnaire in which tolerability, feasibility and satisfaction of VR use is evaluated.
  Arms: VR group

SUMMARY:
SUMMARY

Rationale: The use of an external cephalic version (ECV) to rotate the fetus from a non-cephalic to cephalic presentation reduces the rate of caesarean section by approximately two-thirds in term pregnancies with breech presentation. Reducing pain during external cephalic version can contribute to an increase in success rate and consequently reduce the number of cesarean sections. Literature about the effectivity of virtual reality (VR) on acute pain reduction seems promising.

Objective: The primary objective of this study is to explore the effect of VR on pain during ECV. Secondary objectives are the rate of successful ECV procedures and to explore tolerability, feasibility and patient satisfaction of VR use.

Study design: The study concerns a non-blinded, single centre, randomised controlled trial.

Study population: Eligible women who fulfill the inclusion criteria and are scheduled for an external cephalic version in the Zuyderland Medical Centre location Heerlen.

Intervention: The study population will be randomly divided into the intervention group (VR-group) or the standard care group. The intervention group can choose for an immersive guided relaxation VR experience or an interactive VR experience during the external version additional to the usual standard care. The participants randomised to the standard care group receive the usual standard care given during external version.

Main study parameters/endpoints: The primary outcome is pain measured on a numeric rating scale (NRS). A total of 42 patients have to be included in each group. This means that a total of 84 women will have to be included in the study.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Each participating woman is asked to complete a questionnaire after using VR and the degree of pain perception is questioned on the basis of a 0-10 score (NRS). The study population experiences a very small medical risk when participating to this study. They can experience side-effects of VR for example dizziness or nausea and in rare cases epileptic insults.

ELIGIBILITY:
Inclusion Criteria:

* Written and orally given informed consent
* 18 years and older
* Native Dutch speaker
* Singleton pregnancy in breech position
* Scheduled ECV

Exclusion Criteria:

* Contraindication for ECV
* Chronic pain patients defined as 'persistent or recurrent pain lasting longer than 3 months' [16]. The pain is not due to an obstetrical problem.
* Chronic use of pain medication (opioids)
* Alcohol or drug abuse
* Known car sickness
* Epileptic insults in previous history
* Psychotically seizures in previous history
* Claustrophobic
* Blindness
* History of mental illness
* Patients in strict isolation (MRSA)
* Age <18 years
* Twin pregnancy
* No native Dutch speaker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change of pain during ECV when using VR (VAS, visual analogue scale) | 15 minutes
  pain score by VAS visual analogue scale minimum 0-maximum 10 (higher score is a worse outcome).

SECONDARY OUTCOMES:
Rate of successful ECV procedures | 15 minutes
Patient tolerability, feasibility and satisfaction of VR use (questionnaire) | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: M Wassen, Dr, Principal Investigator — Zuyderland MC
Locations (1):
- Zuyderaland MC, Heerlen, Netherlands